CLINICAL TRIAL: NCT00004114
Title: Non-Myeloablative Chemotherapy Followed by Unrelated Allogeneic Stem Cell Transplantation in Patients With Advanced Hematologic Malignancies: A Pilot Study
Brief Title: Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Advanced Hematologic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study never opened
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067340; UCLA-9902026; NCI-G99-1603
Record Dates: First submitted 1999-12-10; First posted 2004-02-16 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2012-07

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes
Keywords: recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic myelomonocytic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; previously treated myelodysplastic syndromes; AIDS-related peripheral/systemic lymphoma; recurrent mantle cell lymphoma; anaplastic large cell lymphoma; refractory cytopenia with multilineage dysplasia; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelomonocytic, Chronic; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — Filgrastim; Cyclophosphamide; Cytarabine; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: cytarabine
Drug: fludarabine phosphate
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill cancer cells.

PURPOSE: Phase I trial to study the effectiveness of chemotherapy plus peripheral stem cell transplantation in treating patients who have advanced hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of allogeneic engraftment after unrelated matched allogeneic peripheral blood stem cell transplantation preceded by a nonmyeloablative, fludarabine based conditioning regimen in patients with advanced hematologic malignancies. II. Determine the toxicities of this regimen, especially graft versus host disease, in these patients.

OUTLINE: Patients receive fludarabine IV over 30-60 minutes on days -7 to -4, cyclophosphamide IV over 30 minutes on days -7 to -5, and cytarabine IV over 2 hours on days -4 and -3. Allogeneic peripheral blood stem cells are infused on day 0. Filgrastim (G-CSF) is administered IV over 1 hour or subcutaneously beginning on day 1 and continuing until blood counts recover. Patients are followed weekly until day 60 and then monthly for 10 months.

PROJECTED ACCRUAL: A total of 6 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced hematologic malignancy unsuitable for standard allogeneic bone marrow transplantation One of the following types: Refractory or relapsed acute myelogenous or lymphocytic leukemia Over 55 years Chronic myelogenous leukemia and failed interferon treatment Over 55 years Lymphoma, chronic lymphocytic leukemia, Hodgkin's disease, or multiple myeloma: Refractory OR More than 2 relapses OR Relapse after autologous peripheral blood stem cell transplantation Myelodysplastic syndrome other than refractory anemia Severe aplastic anemia Under 55 years and either organ dysfunction or not eligible for standard allogeneic bone marrow transplant due to one or more of the following: Chronic hepatitis LVEF less than 50% Karnofsky less than 70% Unrelated matched donor available

PATIENT CHARACTERISTICS: Age: See Disease Characteristics Adult Performance status: See Disease Characteristics Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: See Disease Characteristics SGOT/SGPT no greater than 4 times upper limit of normal Renal: Creatinine no greater than 2 mg/dL Cardiovascular: See Disease Characteristics Pulmonary: DLCO at least 50% predicted Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Study Chair — Jonsson Comprehensive Cancer Center